CLINICAL TRIAL: NCT00004143
Title: Allogeneic Mixed Chimerism Stem Cell Transplantation Utilizing In Vivo and In Vitro Campath for Hemoglobinopathies and Bone Marrow Failure Syndromes
Brief Title: Allogeneic Mixed Chimerism Stem Cell Transplant Using Campath for Hemoglobinopathies & Bone Marrow Failure Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Rizzieri, MD (Other)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, MD, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008771; DUMC-1340-99-7 (Other: Duke University Medical Center Institutional Review Board); NCI-G99-1617 (Other Grant/Funding Number: National Cancer Institute); CDR0000067374
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Sickle Cell Anemia; Severe Aplastic Anemia; Paroxysmal Nocturnal Hemoglobinuria (PNH); Pure Red Cell Aplasia
Keywords: sickle cell anemia; severe aplastic anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Red-Cell Aplasia, Pure | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Campath SCT for hemoglobinopathies (Experimental): Campath, Chemo and/or TBI Allo SCT
  Interventions: Drug: Campath, Chemo and/or TBI Allo SCT
- Campath SCT for Bone Marrow Failure (Experimental): Campath, Chemo and/or TBI Allo SCT
  Interventions: Drug: Campath, Chemo and/or TBI Allo SCT

INTERVENTIONS:
Drug: Campath, Chemo and/or TBI Allo SCT — Allogeneic PBSC/marrow will be collected/harvested from the donor after granulocyte colony-stimulating factor (G-CSF) priming. The allogeneic PBSCs will be infused as per current institutional practice.
  Other Names: Alemtuzumab; Allogeneic Hematopoietic Stem Cell Transplant

SUMMARY:
RATIONALE: Although used primarily to treat malignant disorders of the blood, allogeneic stem cell transplantation can also cure a variety of non-cancerous, inherited or acquired disorders of the blood. Unfortunately, the conventional approach to allogeneic stem cell transplantation is a risky procedure. For some non-cancerous conditions, the risks of this procedure outweigh the potential benefits. This protocol is designed to test a new approach to allogeneic stem cell transplantation. It is hoped that this approach will be better suited for patients with non-cancerous blood and bone marrow disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective(s):

1. Evaluate the feasibility in terms of mortality, occurrence of acute graft versus host disease, and grades 3-4/4 toxicity of in vivo and in vitro Campath coupled with concomitantly administered nonmyeloablative fludarabine, cyclophosphamide and total body irradiation (TBI) followed by Human Leukocyte Antigen (HLA) 5-6/6 matched family member allo peripheral blood stem cell transplant (PBSCT).
2. Evaluate the engraftment rate of HLA 5-6/6 matched family member patients who receive in vivo Campath followed by concomitantly administered fludarabine, cyclophosphamide and total body irradiation (TBI) as a conditioning regimen with Campath-treated peripheral blood stem cells (in vitro and in vivo exposure).

Secondary Objective(s):

1. Evaluate the response rate and survival of patients who receive a non-myeloablative conditioning regimen of in vivo Campath followed by concomitantly administered fludarabine, cyclophosphamide and total body irradiation (TBI) with Campath-treated peripheral blood stem cells.
2. Evaluate the recovery of immune function post engraftment with this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have their clinical material reviewed at the transplanting institution and the diagnosis confirmed
* Performance status must be Cancer and Leukemia Group B (CALGB) Performance Status (PS) 0, 1, or 2.
* Patients must have a 5/6 to 6/6 HLA matched family member donor who is evaluated and deemed able to provide PBSCs and/or marrow by the transplant team. Donor must have < 50% Hemoglobin S (HgS) on hemoglobin electrophoresis. Cytomegalovirus (CMV) status of the donor will be assessed, but not used as an exclusion criterion.
* Patients must meet the following laboratory parameters unless due to disease status as determined by the treating physician:

  1. bilirubin and hepatic transaminases and creatinine must be reviewed by the transplantation center and deemed acceptable.
  2. HIV antibody negative.
  3. hematocrit, white cell count, platelet counts and hematologic status will be reviewed by the treating physician before patient is deemed acceptable.
* Patient must agree to use some form of adequate birth control during the periods that they receive chemotherapy and any post-chemotherapy medications related to the transplant.
* Patients must also have a resting multiple gated acquisition scan (MUGA) or echocardiogram and Pulmonary Function Tests (PFTs) with Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) performed before transplant. Recommended minimum standards include an Ejection Fraction (EF) greater than 40% and DLCO greater than 40% for this less toxic regimen.
* Appropriate cardiology or pulmonary consultations should be considered if the patient has severe cardiac or lung disease at the initiation of therapy.

I) Hemoglobinopathies:

(a)Sickle Cell Anemia having history of one or more of the following despite treatment with standard therapies such as hydroxyurea: i) 2 or more episodes of acute chest syndrome since age 13 years ii) pulmonary hypertension as measured by tricuspid regurgitant jet velocity of greater than 2.5m/s iii) 2 or more painful crisis per year requiring medical care and analgesia in excess of what is needed at baseline.

iv) history of cerebrovascular accident (b)Thalassemia major: Those eligible will have either cardiac or hepatic sequela of thalassemia as documented by biopsy or functional studies. For those with hepatic damage, this would be an increase in size by 50% of the liver or a doubling of the total bilirubin, aspartate transaminase (AST), alanine aminotransferase (ALT), or alkaline phosphatase. To be eligible for transplant due to cardiac damage, there must be evidence of left ventricular dysfunction as measured by MUGA scan or echocardiography.

II) Bone marrow failure Disorders

1. Severe Aplastic Anemia: Cytopenia consisting of at least 2 of the following 3: absolute neutrophil count less than 500/μL, platelet count less than 20,000/μL, and reticulocyte count less than 50,000/μL.
2. Paroxysmal nocturnal hemoglobinuria (PNH): Patients must have a history of either life-threatening thrombosis, cytopenia, transfusion dependence or recurrent, debilitating hemolytic crisis
3. Pure red cell aplasia: Patients must be transfusion dependent.

Exclusion Criteria:

* pregnant or lactating women,
* patients with other major medical or psychiatric illnesses which the treating or transplant physician feels could seriously compromise compliance to this protocol
* patients with known history of allergies to murine protein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 1999-09; Primary Completion 2008-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Rizzieri, MD, Study Chair — Duke Cancer Institute; Mitchell Horwitz, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Duke Cancer Institute, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was reopened in 2003 for non-malignant conditions only. Enrollment closed in 2008 due to lack of enrollment.
Period: Overall Study
Arm/Group | All Patients
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Neutrophil Engraftment
Description: Number of patients with neutrophil engraftment: Absolute Neutrophil Count (ANC) > 500/μL and hemoglobin level remaining above 10 g/dL without transfusion support, with tests showing at least 2.5% donor cells present. Primary graft failure is defined as absence of establishment of adequate donor hematopoiesis by day 42 with bone marrow cellularity < 5%, peripheral White Blood Count (WBC) < 500/μL, peripheral ANC < 100/μL, and/or platelets < 10,000/μL by day 120 with absence of megakaryocytes in the bone marrow (in the absence of disease relapse).
Time Frame: 1 year post transplant
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 2
participants | 2

2. Primary Outcome: Number of Patients With Platelet Engraftment
Description: Number of patients with platelet engraftment - Platelets > 20,000/μL and hemoglobin level remaining above 10 g/dL without transfusion support, with tests showing at least 2.5% donor cells present. Primary graft failure is defined as absence of establishment of adequate donor hematopoiesis by day 42 with bone marrow cellularity < 5%, peripheral White Blood Count (WBC) < 500/μL, peripheral ANC < 100/μL, and/or platelets < 10,000/μL by day 120 with absence of megakaryocytes in the bone marrow (in the absence of disease relapse).
Time Frame: 1 year post transplant
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 2
participants | 2

3. Secondary Outcome: Overall Survival
Description: Number of patients alive 2 years after transplant
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 2
participants | 2

4. Primary Outcome: Number of Patients With Grade 3-4 Acute Graft Versus Host Disease (GVHD)
Description: Number of patients with Grade 3-4 acute Graft Versus Host Disease (GVHD). GVHD will be monitored at least two times per week through day 45, then weekly through day 60 and graded by 2 persons at each institution, to ensure internal consistency in grading.
Time Frame: 60 days post transplant
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 2
participants | 2

5. Primary Outcome: Number of Participants With Grade 3-4 Unexpected Adverse Events
Description: An unexpected adverse event is one that differs in the nature, severity, or frequency from (a) the research procedures that are described in the protocol-related documents, (such as the IRB-approved research protocol and informed consent document) as expected, and/or (b) the characteristics of the subject population being studied.
Time Frame: 45 days post transplant
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 2
participants | 0

6. Primary Outcome: Number of Participants With Transplant-related Mortality
Description: Number of patients who died due to transplant-related complications
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Time Frame: 45 days post transplant
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=2)
Hypertension (Cardiac disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Cardiac ischemia / infarction (Cardiac disorders) | 1 (1)
Parainfluenza (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No